CLINICAL TRIAL: NCT01409876
Title: HistoScanning- Based Dose-painting Image-guided Interstitial PDR-brachytherapy in Prostate Cancer - a Phase II Trial
Brief Title: HistScanning- Based PDR Brachytherapy in Prostate Cancer HistoScanning- Based Interstitial PDR Brachytherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Sebastian Lettmaier, University Hospital Erlangen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HistoBrachy1
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: histoscanning; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

ARMS (1):
- Brachytherapy (Experimental)
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — interstitial image- guided PDR/HDR brachytherapy

SUMMARY:
This is a phase II trial looking at the feasibility of HistoScanning- based dose-painting image- guided interstitial brachytherapy in non- metastatic prostate cancer

Endpoints:

Primary endpoint Evaluation of the feasibility of HistoScanning- based dose-painting image- guided interstitial brachytherapy

Secondary endpoints

1. Evaluating tumor response using HistoScanning
2. Evaluating locoregional recurrence rates by measuring PSA
3. Analysis of the correlation between tumor response as determined by HistoScanning and PSA response
4. Evaluating the safety dose-painting image- guided interstitial brachytherapy by recording serious adverse events

DETAILED DESCRIPTION:
Rationale:

The study is designed as a prospective monocentric phase II trial. The choice of the therapeutic concept is governed by the risk group that the patient falls into. Risk groups are defined according to the classification by D' Amico.

The following concepts will be used:

HDR brachytherapy: 19,0- 38 Gy / 2-4 fractions (2-4 x 9,5 Gy)

PDR brachytherapy: 35-70 Gy / 50 --100 pulses(1 puls/h, 24 h/d)

Dose painting the timorous areas as seen in HistoScanning as covered with a dose Dref2>130-150%

External beam radiotherapy will be used in addition to brachytherapy for intermediate and high risk patients. The following concepts will be used 50,40 Gy / 28 fractions at 1.8 Gy

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer
* All cT1-3 carcinomas independent of grading and PSA value
* Prostate volume< 70cc
* No distant metastases
* Karnofsky > 60
* Written informed consent from the patient regarding study participation

Exclusion criteria:

* All patients who do not meet the inclusion criteria
* T4 carcinomas
* Proven metastases N+ and/or M1
* Epidural or general anaesthesia not possible
* Pathological clotting parameters

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the feasibilty of histoscanning- based dose-painting image- guided interstitial brachytherapy | 5 years

SECONDARY OUTCOMES:
assessing tumor response and side effects | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Therapy University Hospital, Erlangen, Germany

REFERENCES:
- [Derived] Strnad V, Lotter M, Kreppner S, Fietkau R. Brachytherapy focal dose escalation using ultrasound based tissue characterization by patients with non-metastatic prostate cancer: Five-year results from single-center phase 2 trial. Brachytherapy. 2022 Jul-Aug;21(4):415-423. doi: 10.1016/j.brachy.2022.02.003. Epub 2022 Apr 6. PMID 35396138